CLINICAL TRIAL: NCT03628027
Title: The Antidepressant Advisor: A Decision Support System for UK Primary care-a Feasibility Study
Brief Title: The Antidepressant Advisor Study
Acronym: ADeSS
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: King's College London (Other)
Collaborators: NHS Lambeth Clinical Commissioning Group (Other); EMIS PLC (Unknown); D'Or Institute for Research and Education (Other)
Responsible Party: Principal Investigator, Dr Roland Zahn, Senior Clinical Lecturer, Honorary Consultant Psychiatrist, King's College London
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: PB-PG-0416-20039
Record Dates: First submitted 2018-08-01; First posted 2018-08-14 (Actual); Last update posted 2020-07-30 (Actual); Status verified 2020-07

CONDITIONS: Major Depressive Disorder
Keywords: Major Depressive Disorder; Antidepressant Medication; Digital Health; Computerised Decision Support Tool
MeSH Terms: conditions — Depressive Disorder, Major

STUDY DESIGN:
Intervention Model Description: Cluster-randomised controlled clinical trial. GPs are randomised in blocks of N = 2 to a treatment arm. All patients under the care of a GP receive the treatment to which the GP was randomised.
Who Masked: Participant, Outcomes Assessor
Masking Description: GPs will need to be made aware of their treatment arm in order to implement the correct treatment. However, this should not be disclosed to patients, either by the GP or Trial Co-ordinator who will also be blinded.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Treatment Algorithm (Experimental): The treatment algorithm arm will be the experimental arm in which GPs use the computerised decision support tool to guide their prescribing of antidepressants.
  Interventions: Device: Computerised decision support algorithm
- Treatment-as-usual (No Intervention): The treatment-as-usual arm will comprise GPs prescribing antidepressants and providing care as they typically would.

INTERVENTIONS:
Device: Computerised decision support algorithm — The algorithm is integrated into the EMIS computer system used by GPs. The algorithm advises on which antidepressants should be prescribed based on a patient's treatment history.
  Arms: Treatment Algorithm

SUMMARY:
The Antidepressant Advisor Study is a feasibility study to develop and probe the feasibility of a computerised decision support tool for GPs to prescribe antidepressant treatments. The study will use an algorithm to support GPs in their prescribing decisions for patients who have previously not responded to first-line antidepressants. Another group of GPs will prescribe as usual without the algorithm so that the effectiveness of the tool can be assessed, in terms of patient recovery. The aim of the study is to design a support tool which can aid GPs to prescribe the most effective treatment option for the patient so that they have increased likelihood of improvement in depression. A further aim of the study is to assess GP adherence and satisfaction with the tool so that modifications can be made that would improve the usability of the tool in future trials.

DETAILED DESCRIPTION:
To address the urgent need for user-friendly decision support for antidepressant choices in UK primary care, the investigators will probe a specifically tailored innovative tool advising GPs on patients who have not responded to first-line treatments. Despite one promising US study, there is no such tool available in the UK. The US study was based in a private GP setting and employed now outdated treatment algorithms. In contrast, the treatment algorithm implemented in the current decision support tool is based on National Institute for Health and Care Excellence (NICE) guidelines including the latest health technology appraisals. The investigators have further gained the support of the leading UK provider of primary care electronic record systems (EMIS group: >3000 GP practice users) who will develop the software implementation of the algorithm as an add-on tool to their widely employed software.

Considering complex intervention guidance, the study is designed as a feasibility study to provide estimates of the following unknown variables needed to plan a subsequent larger trial: lost to follow-up and recruitment rates, GP satisfaction with the tool, impact on health service use, and standard deviations on our planned primary outcome measure on the self-rated Quick Inventory of Depressive Symptomatology (QIDS-SR16) for a subsequent trial. The investigators will use a single-blinded parallel group cluster-randomised controlled trial design with at least 8 GPs across 8 practices (one per practice) being randomised supported by the Clinical Research Network (CRN) to two arms: 1) Usual care of patients with depression with no computerised decision support, 2) Using the novel computerised decision support tool to assist with antidepressant choices.

The investigators will recruit 8-20 GPs in 8-20 different practices to avoid communication between GPs, each contributing approximately 10 study patients. The EMIS eligibility tool (see below) will identify potential participants by screening for antidepressant and problem history. Blinded practice staff/CRN will ask all eligible patients for consent for contact. Patients will fill in an electronic version of the self-report version of the Primary Care Evaluation of Mental Disorders (PRIME-MD) and provide electronic consent for this. Alternatively, participants will be called to answer the questions over the phone and provide oral consent. Other patients will prefer receiving a mailed printed questionnaire and provide written consent. PRIME-MD has been validated against clinical diagnoses of current major depressive and anxiety disorders, as well as alcohol abuse according to DSM-IV criteria and will be modified to screen for drug abuse and anxiety disorders may be dropped from the screening as they are not exclusion criteria and will be assessed in the in-depth assessment. Patients will further complete self-report versions of the WHO Composite International Diagnostic Interview (CIDI) screening scale for bipolar disorder and 3 screening questions validated in the investigators' group to exclude schizophrenia. Further, the investigators will ask about the inclusion and exclusion criteria for the study, because the information recorded on EMIS is not always complete and does not always include a patient's history with previous GP surgery for example. Eligible patients will be seen for an in-depth assessment by the study research associate (RA) where she will take written informed consent.

2.1.2 Data collection and Assessment for patients meeting the pre-screening criteria

As in the investigators' previous work, the RA will be closely supervised and trained, establishing sufficient inter-rater reliability on semi-structured interviews with the PI before carrying out assessments independently. Apart from the outcome measures, the in-depth assessment will include measuring past subthreshold hypomanic symptoms, and perceived credibility of and expectancy towards treatment using a dedicated questionnaire, and a detailed clinical evaluation whilst accessing patients' EMIS records including:

* Treatment history
* Medical history
* Age at onset, episode duration and number, illness duration
* International Neuropsychiatric Interview (MINI) suicidality screen
* DSM5 Structured Clinical Diagnostic Interview
* Addenbrooke's Cognitive Examination-R in patients over 50 to detect early Alzheimer's disease
* Young Mania Rating Scale The results of the assessment will be shared with GPs and patients. This will also allow the investigators to use the Maudsley Staging Method to compare the level of treatment resistance between treatment groups prior to entry into the study as a potential confounder. Patients who meet the inclusion/exclusion criteria will subsequently be seen by their GP who initiates and monitors treatment using EMIS. The decision whom to include will not be made by the GPs to ensure against different selection biases in the different treatment arms. The RA will be blinded to the intervention arm that a GP was randomised to, in order to prevent the RA from making biased inclusion/exclusion decisions. The RA will communicate inclusion/exclusion decisions to patients and will draft a short report to their GP. The RA will seek the Chief Investigator's advice on inclusion/exclusion questions without telling him which GP the patient was referred from. Should the RA become unblinded accidentally or for some other reason, this would be noted in the case record file, but the patient would be retained in the study. On the second and final RA visit 15-18 weeks after the baseline assessment, outcome measures and Young Mania Rating Scale will be repeated and the Longitudinal Interval Follow-up Interview will be used to determine remission, its psychiatric status rating scale will be used at baseline for comparison. After being enrolled, patients, who have no smartphone, receive a mobile smart phone to access a secure patient app (developed as part of the proposal which will communicate via secure email with GPs) to prompt them to enter weekly (changing the usual two week time interval to one week and using the Maudsley modified version) PHQ-9 ratings (chosen also because it has no licencing restrictions), to report hypomanic symptoms, fill in a validated self-report side effects scale (Frequency, Intensity, and Burden of Side Effects Rating (FIBSER), and enter medication (including opting in for a reminder function), as well as asking about self-blame-related action tendencies such as hiding. The app will be based on an adaptation of similar mood tracking apps developed by our BRC. Alternatively, ratings and medication compliances will be asked about at weekly intervals via post or phone which will be recorded in the case file.

Main objectives of this study

1. To develop the first computerised decision support tool for antidepressant treatment in UK primary care
2. To probe the feasibility of a clinical trial to assess the tool's efficacy by

   1. estimating lost to follow-up rates
   2. estimating GP and patient adherence to prescribed medications
   3. determining the number of GP practices willing to recruit patients for the study (determined by the CRN who will approach all practices in the participating CCGs)
   4. estimating the recruitment rates per GP
   5. estimating GP satisfaction
3. To provide standard deviation estimates and intra-class correlation coefficients per GP for computing effect size estimates for improving treatment outcomes in preparation of larger subsequent trials
4. To collect health economic estimates of changes in service use associated with the new tool (including psychiatric referrals to mental health teams and/or the study psychiatrist).

As soon as possible after their baseline in-depth assessment, eligible patients will undergo treatment over 14 weeks with their GPs which allows 3 weeks for determining sufficient treatment response at low and high dose of each of the two different recommended medications and 1 week for cross-tapering before step 1 and step 3. The final assessment by the RA will take place 15-18 weeks after the baseline assessment. Patients' participation will therefore last for approximately 15-18 weeks. Deviations from this time will occur due to scheduling difficulties and will be recorded. Time in the study will be used as a covariate in secondary data analyses.

GPs will be randomised into two groups, asking each GP to enroll approximately 8-11 participants each, adding more GPs if necessary. The study aims to recruit 86 participants assuming the same lost to follow-up rate as in the US trial (18%), resulting in a final sample size of 70 (35 in each group as recommended). This will enable the investigators to estimate the lost to follow-up rate within a 95% confidence interval of +/-8%. Because the comparable previous trial did not provide effect size estimates, this study has been designed to provide means and standard deviations, as well as confidence intervals for measures of change on the primary outcome measure (QIDS-SR16) in n=35 per group as recommended for feasibility trials.

Double data entry will be employed. Categorical outcomes (e.g. lost to follow-up rate) will be described using appropriate summary statistics. The QIDS-SR16 and other continuous outcomes will be summarised at baseline and final assessment time points to obtain means and standard deviations for a larger trial sample size calculation, with the GP intra-class correlation calculated for the outcome variable using one-way random effects analysis of covariance (adjusted for baseline). The investigators plan to do a preliminary analysis of the difference between the groups, as far as possible using the intention to treat principle. This analysis will be identified as preliminary and underpowered when published. The outcomes measured at baseline and follow-up only, such as the QIDS-SR16, will be analysed using robust linear regression to account for clustering within GP. Continuous outcomes measured weekly will be analysed using mixed linear regression models with an intercept for GP to account for clustering. Both types of models will include treatment group as a covariate, in order to estimate differences between the two intervention groups, and will adjust for the baseline measure of the outcome where appropriate. The investigators do not expect missing baseline data, however, any such missing data will be imputed using mean imputation. Missing data in the weekly outcomes will be accounted for under the missing at random assumption by using the maximum likelihood algorithm to fit the mixed models. The investigators may consider multiple imputation for outcomes measured only at follow-up if post-randomisation adherence variables can be quantified and are related to having missing outcomes.

ELIGIBILITY:
Inclusion Criteria:

* age 18 years +
* at least moderately severe major depressive syndrome on PHQ-9 (score 15 +)
* no plans to change GP practice
* able to complete self-report scales orally or in writing
* no previous prescription of mirtazapine or vortioxetine
* early treatment resistance as defined by 1) current or recent prescription (in the last 2 months) of any of the following antidepressants: citalopram, fluoxetine, sertraline, escitalopram, paroxetine, venlafaxine, or duloxetine AND 2) previous prescription of at least one other antidepressant out of the same list.

Exclusion Criteria:

* inability to consent to study
* unstable medical condition
* currently receiving specialist psychiatric treatment
* high suicide risk (MINI suicidality screen)
* past diagnosis of schizophrenia or schizo-affective disorder
* current psychotic symptoms (3 clinical screening questions)
* bipolar disorder
* currently at risk of being violent
* drug (modified PHQ) or alcohol abuse (PHQ) over last 6 months
* suspected central neurological condition
* pregnancy or insufficient contraception in women of childbearing age
* breastfeeding or within 6 months of giving birth in women of childbearing age
* both escitalopram and sertraline have already been prescribed

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 86 (Estimated)
Dates: Start 2018-08-01 (Actual); Primary Completion 2021-04 (Estimated); Study Completion 2021-07 (Estimated)

PRIMARY OUTCOMES:
Self-Rated Quick Inventory of Depressive Symptomatology (QIDS-SR16) | 16 weeks
  Change from baseline depressive symptoms (not primary outcome for this feasibility study, only for full trial, primary feasibility outcomes are listed from 6 onwards). Total scale range: 0 - 48. Higher score indicates more change in depressive symptoms.

SECONDARY OUTCOMES:
Montgomery Asberg Depression Rating Scale (MADRS) | 16 weeks
  Change from baseline depressive symptoms. Total scale range: 0 - 60. Higher score indicates more change in depressive symptoms.
Clinical Global Impression | 16 weeks
  Change from baseline severity Total scale range: 1 - 7. Lower score indicates more improvement in symptoms.
Generalised Anxiety Disorder (GAD-7) | 16 weeks
  Change from baseline anxiety symptoms used in the NHS. Total scale range: 0 - 21. Higher score indicates more change in anxiety symptoms.
Body Mass Index (BMI) | 16 weeks
  Change from baseline healthy weight. Total range: 12 - 42. Higher score indicates more change in BMI.

OTHER OUTCOMES:
Recruitment Rate | Through study completion, an average of 16 months
  Rate at which patients are recruited to the study
Lost to Follow-up Rate | Through study completion, an average of 16 months
  Rate at which patients are lost to follow-up
Adverse Event Rate | Through study completion, an average of 16 months
  Grade and rate at which adverse events occur
Helpfulness, ease of use and workload of intervention using King's GP Satisfaction Measure | Through study completion, an average of 16 months
  Average GP satisfaction. Includes recommendation for future clinical use, and opinion on usefulness to patient care. Subscale ranges-Q1: 0 - 11, Q2: 0 - 6 (higher score indicates more improved care), Q3: 0 - 6 (higher score indicates higher workload), Q4: 0 - 6 (higher score indicates higher helpfulness), Q5: 0 - 6 (higher score indicates higher workload), Q6: 0 - 6 (higher score indicates easier to use), Q7: 0 - 6 (higher score indicates more improvement in care), Q8: 0 - 6 (higher score indicates better than other tools), Q9: 0 - 6 (higher score indicates less likelihood to ignore tool), Q10: 0 - 6 (higher score indicates more strongly recommend)
GP Adherence to Algorithm | Week 16
  Assessed for each patient by trial clinician, from 0 (none of the recommended steps implemented) to 3 (fully implemented)
Service Use (EMIS) | Week 16
  Information taken from EMIS, including psychiatric referrals, referrals to study psychiatrist, time to psychiatric referral
Adult Service Use Schedule (AD-SUS) | Week 16
  Assessed on routine validated KCL questionnaire. Subscale ranges: Q1: 0 (no) 1 (yes), Q2: continuous number, Q3: 0 (no), 1 ( yes), Q4: continuous number, Q5: 0 (no), 1 (yes), Q6: text answer, Q7: continuous number
Euroqol Quality of Life Measure (EQ-5D-3L) | Week 16
  Change from baseline quality of life. Assessment of cost-effectiveness of intervention. Visual analogue question range: 0 - 100. Higher score indicates better perceived health.
Average % Patient Adherence (EMIS) | Week 16
  Information taking from EMIS including prescribing records
Social and Occupational Functioning Assessment Scale (SOFAS; DSM-V) | Week 16
  Change from baseline psychological functioning
Maudsley Visual Analogue Mood Scale | Week 16
  Change from baseline mood. Total scale range: 0 - 300. Higher scores indicate more improvement in mood.
Patient Adherence | Week 16
  Information taken from EMIS including % of attended GP visits out of total scheduled number
Frequency, Intensity and Burden of Side Effects Rating (FIBSER) | Weekly for 16 weeks
  Average score for medication side effects. Each subscale range: 0 - 6. Higher scores indicate more burdensome side effects.
Average % Patient Adherence (Mobile App) | Weekly for 16 weeks
  Adherence to prescribed antidepressants
Average Maudsley Modified Patient Health Questionnaire (PHQ-9) | Weekly for 16 weeks
  Average depression score over last 2 weeks. Total scale range: 0 - 21. Higher scores indicate more depressive symptoms.

CONTACTS AND LOCATIONS:
Overall Officials: Roland Zahn, Principal Investigator — Senior Clinical Lecturer, Honorary Consultant Psychiatrist
Locations (1):
- King's College London, IoPPN, London, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] NICE. Depression: The treatment and management of depression in adults. The British Psychological Society and The Royal College of Psychiatrists; 2010.
- [Background] Symons L, Tylee A, Mann A, Jones R, Plummer S, Walker M, Duff C, Holt R. Improving access to depression care: descriptive report of a multidisciplinary primary care pilot service. Br J Gen Pract. 2004 Sep;54(506):679-83. PMID 15353054
- [Background] Kurian BT, Trivedi MH, Grannemann BD, Claassen CA, Daly EJ, Sunderajan P. A computerized decision support system for depression in primary care. Prim Care Companion J Clin Psychiatry. 2009;11(4):140-6. doi: 10.4088/PCC.08m00687. PMID 19750065
- [Background] Rollman BL, Hanusa BH, Lowe HJ, Gilbert T, Kapoor WN, Schulberg HC. A randomized trial using computerized decision support to improve treatment of major depression in primary care. J Gen Intern Med. 2002 Jul;17(7):493-503. doi: 10.1046/j.1525-1497.2002.10421.x. PMID 12133139
- [Background] Lythe KE, Moll J, Gethin JA, Workman CI, Green S, Lambon Ralph MA, Deakin JF, Zahn R. Self-blame-Selective Hyperconnectivity Between Anterior Temporal and Subgenual Cortices and Prediction of Recurrent Depressive Episodes. JAMA Psychiatry. 2015 Nov;72(11):1119-26. doi: 10.1001/jamapsychiatry.2015.1813. PMID 26445229
- [Derived] Harrison P, Carr E, Goldsmith K, Young A, Ashworth M, Fennema D, Duan S, Barrett BM, Zahn R. Antidepressant Advisor (ADeSS): a decision support system for antidepressant treatment for depression in UK primary care - a feasibility study. BMJ Open. 2023 Mar 3;13(3):e060516. doi: 10.1136/bmjopen-2021-060516. PMID 36868594
- [Derived] Harrison P, Carr E, Goldsmith K, Young AH, Ashworth M, Fennema D, Barrett B, Zahn R. Study protocol for the antidepressant advisor (ADeSS): a decision support system for antidepressant treatment for depression in UK primary care: a feasibility study. BMJ Open. 2020 May 24;10(5):e035905. doi: 10.1136/bmjopen-2019-035905. PMID 32448796